CLINICAL TRIAL: NCT06089187
Title: A Comparative Analysis of Elevated Endotracheal Tube Cuff Pressure Incidence in Elective Laparoscopic Abdominal Surgery: Saline vs. Air Inflation
Brief Title: Comparing Endotracheal Tube Cuff Pressure in Laparoscopic Abdominal Surgery: Saline vs. Air Inflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Principal investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETTSVA
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Air; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline Group (Active Comparator): Anesthesia machine's APL valve will be adjusted to a pressure of 20 cmH20, and during ventilation with a balloon, the endotracheal tube cuffs will be inflated with saline in such a way that there will be no leakage sound from the patient's mouth.
  Interventions: Procedure: Endotracheal intubation using an endotracheal tube with cuff inflated with saline
- Air Group (Placebo Comparator): Anesthesia machine's APL valve will be adjusted to a pressure of 20 cmH20, and during ventilation with a balloon, the endotracheal tube cuffs will be inflated with air in such a way that there will be no leakage sound from the patient's mouth.
  Interventions: Procedure: Endotracheal intubation using an endotracheal tube with cuff inflated with air

INTERVENTIONS:
Procedure: Endotracheal intubation using an endotracheal tube with cuff inflated with air — After endotracheal intubation, the endotracheal tube cuff is inflated with air
  Arms: Air Group
Procedure: Endotracheal intubation using an endotracheal tube with cuff inflated with saline — After endotracheal intubation, the endotracheal tube cuff is inflated with saline
  Arms: Saline Group

SUMMARY:
In this study, the investigators aim to compare the incidence of cuff pressure increase between endotracheal tubes inflated with air or saline during elective laparoscopic abdominal surgery under general anesthesia with N2O. This prospective observational study will be conducted on 60 patients aged 18-65 with ASA physical status I-II undergoing elective laparoscopic abdominal surgery under general anesthesia. Patients are randomly assigned to two groups: one group has tubes inflated with air (Group H, n=30), while the other group has tubes inflated with saline (Group S, n=30). The cuff pressure is continuously monitored using a pressure transducer attached to the cuff via a three-way tap. Anesthesia maintenance is achieved with sevoflurane and oxygen/N2O (%40/%60) in both groups. The intervention is performed whenever the cuff pressure exceeds 20 mmHg for >30 seconds during the CO2 insufflation of the abdomen, and the pressure is reduced. The number of interventions is recorded as the primary outcome of the study. The cuff pressure is measured before and after insufflation and after the patients are placed in Trendelenburg and reverse Trendelenburg positions.

DETAILED DESCRIPTION:
The study is designed as prospective and observational research, which takes place at the Balcalı Hospital of Çukurova University between July 2023 and October 2023. After obtaining written informed consent from the participants and approval from the Çukurova University Clinical Research Ethics Committee (Date: 13.07.2023 and Decision no: 186/10), a total of 60 patients, aged between 18-65, with ASA 1-2 risk category, and expected surgical duration of 30-120 minutes, are included in the study for elective laparoscopic abdominal surgery. The exclusion criteria include neuropsychiatric diseases, muscle diseases, significant cardiovascular and respiratory system diseases, upper respiratory tract infection within the past 14 days, morbid obesity, alcohol or substance dependence, history of bronchospasm, expected difficult intubation, history of tracheostomy, and laryngeal diseases or surgery. After informing the patients about the procedure and obtaining written consent, intravenous (IV) access is established in the preoperative preparation room after an 8-hour fasting period. No premedication is administered. Once the patients are transferred to the operating room, standard anesthesia monitoring including electrocardiography (ECG), non-invasive blood pressure, peripheral oxygen saturation (SpO2), and end-tidal CO2 (EtCO2) are applied. Following 3 minutes of preoxygenation with 100% oxygen, anesthesia induction is performed with a 2 mg/kg IV propofol. TOF (train-of-four) monitor calibration is performed to assess the level of muscle relaxation. Subsequently, 0.6 mg/kg of rocuronium IV is administered for neuromuscular blockade. Fentanyl 1 mcg/kg IV is given during anesthesia induction. Endotracheal intubation (ETI) is performed using a high-volume, low-pressure cuffed endotracheal tube (ETT) with an internal diameter of 7-7.5 mm for female patients and 8-8.5 mm for male patients, once the TOF measurement reaches 0. The intubation procedure is carried out by an experienced anesthesiologist using a Macintosh laryngoscope. According to the randomization table created with a computer program, patients who are randomly selected after endotracheal intubation have the APL valve of the anesthesia machine adjusted to a pressure of 20 cmH20, ensuring that there is no air leakage sound from the patient's mouth during ventilation. The ETT cuffs of patients in Group H are inflated with air, while those in Group S are inflated with saline. The cuff pressure is continuously monitored using a pressure transducer connected to the cuff balloon through a three-way stopcock. The transducer set is filled with saline to ensure no air is present. It is connected to a three-way stopcock at the desired measurement point level. All connections are taped to prevent disconnection and leaks, and a "For Respiratory Use Only" label is affixed to enhance patient safety. The pressure calibration on the patient monitor is adjusted according to the sternal notch level of the patient, and the cuff pressure value is measured in mmHg. After ETT placement, ventilation of the patient is set as volume-controlled ventilation with a tidal volume of 6-8 ml/kg, frequency of 10-12/min, and EtCO2 of 35-45 mmHg. An esophageal temperature measurement probe is placed to monitor body temperature. Maintenance of anesthesia for all patients is achieved using a gas mixture of sevoflurane and oxygen/nitrous oxide (40%/60%). When the TOF value is 2 during the maintenance of muscle relaxation, rocuronium 0.15 mg/kg is administered intravenously. Nasogastric tubes are placed in all patients. 45 minutes before the completion of the surgery, tramadol 2 mg/kg IV and paracetamol 1 g IV are administered to provide postoperative analgesia. In cases where the intracuff pressure exceeds 20 mmHg for more than 30 seconds during CO2 insufflation, intervention is performed using a three-way stopcock and syringe to reduce the pressure to 18 mmHg, and the number of interventions is recorded. The highest intracuff pressure, ventilator peak pressure, plateau pressure, and PEEP are recorded every 15 minutes during the first minute after CO2 insufflation. In cases where the intracuff pressure exceeds 20 mmHg for more than 30 seconds during this period, intervention is performed to reduce the pressure to 18 mmHg using a three-way stopcock and syringe. The number of interventions is recorded. Additionally, the intracuff pressures before and after the patients are placed in the reverse Trendelenburg and Trendelenburg positions are recorded. At the end of the surgery, 0.04 mg/kg neostigmine IV and 0.01 mg/kg atropine IV are administered to reverse the effects of muscle relaxation. The patients are extubated when they respond adequately to verbal stimuli and the train-of-four (TOF) value is 90% or above. Once sufficient muscle strength and airway safety are ensured, the patients are transferred from the operating room to the postoperative recovery unit.

In our pilot study, we observed that the total number of interventions 30 minutes after insufflation differed significantly between the saline group (mean = 2.31) and the air group (mean = 4.01), with a standard deviation of 1.68. To ensure a 95% power and a significance level of 0.05%, we determined that a sample size of 27 patients per group (total of 57 patients) was necessary. To account for potential data loss, we included 60 patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65,
* American Society of Anesthesiologists physical status 1 or 2
* Expected surgery time of 30-120 minutes,
* Scheduled for elective laparoscopic abdominal surgery

Exclusion Criteria:

* neuropsychiatric disease
* muscle disease
* serious cardiovascular and respiratory system disease
* upper respiratory tract infection in the last 14 days
* morbid obesity
* alcohol or substance addiction
* history of bronchospasm
* expectation of difficult intubation
* history of tracheostomy
* history of laryngeal disease or surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
The number of intervention | 15 minutes
  The number of interventions required to correct intracuff pressure

SECONDARY OUTCOMES:
Peak Airway pressure | 15 minutes
  Peak airway pressure during the intraoperative period is measured in cmH2O.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong J, Jenner P, Poulose S, Moppett IK. The effect of saline versus air for cuff inflation on the incidence of high intra-cuff pressure in paediatric MicroCuff(R) tracheal tubes: a randomised controlled trial. Anaesthesia. 2021 Nov;76(11):1504-1510. doi: 10.1111/anae.15493. Epub 2021 Apr 23. PMID 33891328